CLINICAL TRIAL: NCT05487040
Title: A PHASE 1, OPEN-LABEL, NON-RANDOMIZED STUDY TO INVESTIGATE THE SAFETY AND PK FOLLOWING MULTIPLE ORAL DOSES OF PF-07321332 (NIRMATRELVIR)/RITONAVIR IN ADULT PARTICIPANTS WITH COVID-19 AND SEVERE RENAL IMPAIRMENT EITHER ON HEMODIALYSIS OR NOT ON HEMODIALYSIS
Brief Title: A Study to Measure the Amount of Study Medicine in Blood in Adult Participants With COVID-19 and Severe Kidney Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision to terminate study was due to slow enrolment and FDA input that available data may be enough for dosing recommendations for severe renal disease (subject to review by FDA).
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C4671028; EPIC-SRI (Other: Alias Study Number); 2023-503870-19 (EudraCT Number)
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
Keywords: Severe acute respiratory syndrome coronavirus 2 (SARS-Cov-2); kidney disease; kidney failure; renal disease; renal failure; dialysis; renal dialysis; hemodialysis; coronavirus disease 2019 (COVID-19); COVID; Paxlovid; antiviral; nirmatrelvir; mild to moderate COVID-19; high risk
MeSH Terms: conditions — COVID-19; Kidney Diseases; Renal Insufficiency | interventions — nirmatrelvir; nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-07321332 (nirmatrelvir)/ritonavir participants with severe renal impairment on hemodialysis (Experimental): Patients with Covid-19 infection and severe renal impairment. Capsule and tablet once a day by mouth.
  Interventions: Drug: PF-07321332 (nirmatrelvir)/ritonavir
- PF-07321332 (nirmatrelvir)/ritonavir participants with severe renal impairment not on hemodialysis (Experimental): Patients with Covid-19 infection and severe renal impairment. Capsule and tablet once a day by mouth.
  Interventions: Drug: PF-07321332 (nirmatrelvir)/ritonavir

INTERVENTIONS:
Drug: PF-07321332 (nirmatrelvir)/ritonavir — Patients with Covid-19 infection and severe renal impairment. Capsule and tablet once a day by mouth.
  Other Names: Paxlovid

SUMMARY:
The purpose of this study is to learn about the side effects (safety) of the study medicine PF-07321332 (nirmatrelvir)/ritonavir for the treatment of mild to moderate COVID-19 infection in adults with severe renal impairment. The study will also look at the amounts of study drug in your blood. There will be 24 participants in this study; 12 of them will have severe renal impairment and not be on hemodialysis and 12 of them will be on hemodialysis.

All participants in this study will take PF-07321332 (nirmatrelvir)/ritonavir by mouth for 5 days. During this time, they will have to collect blood samples to measure the study drug levels in their blood. After taking the study drug for 5 days, the participants will have follow-up visits for about another 28 days for a total of about 34 days in the study. The study team will check how each participant is doing during regular visits at the study clinic.

ELIGIBILITY:
Inclusion Criteria:

* Covid-19 infection
* Severe kidney disease (on hemodialysis or not on hemodialysis)

Exclusion Criteria:

* Hospitalized
* Take medications that are not allowed
* Renal transplant patients
* HIV infection

This is not a complete list. Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (52):
- United States (52):
  - Fresenius Kidney Care Huntsville, Huntsville, Alabama
  - Fresenius Kidney Care Rocket City, Huntsville, Alabama
  - Apogee Clinical Research, LLC, Huntsville, Alabama
  - Nephrology Consultants, Huntsville, Alabama
  - Fresenius Kidney Care Chase, Huntsville, Alabama
  - Fresenius Kidney Care Endeavour, Huntsville, Alabama
  - Fresenius Kidney Care Parkway, Huntsville, Alabama
  - Amicis Research Center - Granada Hills, Granada Hills, California
  - Amicis Research Center, Granada Hills, California
  - DaVita Inglewood Dialysis, Inglewood, California
  - Northridge Kidney Center, Northridge, California
  - Clinnova Research - Redondo Beach, Redondo Beach, California
  - Santa Clarita Dialysis, Santa Clarita, California
  - laurel Canyon Dialysis, Sun Valley, California
  - Desert Cities Diaylsis, Victorville, California
  - Desert Cities Dialysis - Hesperia, Victorville, California
  - Fresenius Kidney Care Ft Lauderdale #2036, Fort Lauderdale, Florida
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - Fresenius Kidney Care Florida Kidney Center #1095, Lauderhill, Florida
  - GCP Research, Global Clinical professionals, St. Petersburg, Florida
  - Fresenius Kidney Care Tamarac-JV #6606, Tamarac, Florida
  - Fresenius Kidney Care Hillsborough #100706, Tampa, Florida
  - Genesis Clinical Research, LLC, Tampa, Florida
  - Fresenius Kidney Care Tampa #1130, Tampa, Florida
  - Fresenius Kidney Care Ybor City #1863, Tampa, Florida
  - Fresenius Kidney Care Town and Country #100474, Tampa, Florida
  - Fresenius Kidney Care Carrollwood #1805, Tampa, Florida
  - Fresenius Kidney Care-Boise, Boise, Idaho
  - Fresenius Kidney Care- Caldwell, Caldwell, Idaho
  - Fresenius Kidney Care-Meridian, Meridian, Idaho
  - Liberty Dialysis- Nampa, Nampa, Idaho
  - Boise Kidney & Hypertension Institute, PLLC, Nampa, Idaho
  - Swedish Covenant Hospital, Chicago, Illinois
  - NorthShore University HealthSystem - Evanston Hospital, Evanston, Illinois
  - DaVita Evanston Renal Center, Evanston, Illinois
  - DaVita Glen Dialysis, Glenview, Illinois
  - NorthShore University HealthSystem - Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem - Highland Park Hospital, Highland Park, Illinois
  - NorthShore University HealthSystem - Skokie Hospital, Skokie, Illinois
  - NorthShore Immediate Care Center - Skokie at Old Orchard Woods, Skokie, Illinois
  - NorthShore University HealthSystem - Clinical Trials Center, Skokie, Illinois
  - Piedmont Dialysis Center, Winston-Salem, North Carolina
  - Brookview Hills Research Associates, Winston-Salem, North Carolina
  - Northside Dialysis Center, Winston-Salem, North Carolina
  - Fresenius Kidney Care / Roane County #2829, Harriman, Tennessee
  - Fresenius Kidney Care / Fort Sanders #1597, Knoxville, Tennessee
  - Fresenius Kidney Care / Cedar Bluff #6942, Knoxville, Tennessee
  - Knoxville Kidney Center, PLLC, Knoxville, Tennessee
  - Arlington Nephrology, Arlington, Texas
  - South Arlington Dialysis Center, Arlington, Texas
  - Grand Prairie Dialysis Center, Grand Prairie, Texas
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671028

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated early following completion of Cohort 2. The decision to terminate was not due to safety, but was based on an assessment that available pharmacokinetic (PK) and safety data are sufficient to inform dosing recommendations for participants with severe renal impairment (SRI).
Groups:
- Cohort 1 (No HD): Participants in Cohort 1 had SRI (defined as estimated glomerular filtration [eGFR] rate < 30 milliliter per minute per 1.73 square meter [mL/min/1.73m^2]) not on hemodialysis (HD) and mild to moderate COVID-19 disease with confirmed SARS-CoV-2 infection and initial onset of signs/symptoms attributable to COVID-19 within 5 days prior to the day of treatment assignment. All eligible participants were assigned to receive a single dose of PF-07321332 (nirmatrelvir)/ritonavir 300 mg/100 mg orally on Day 1 followed by PF-07321332 (nirmatrelvir)/ritonavir 150 mg/100 mg once daily (QD) from Day 2 to Day 5.
- Cohort 2 (Intermittent HD): Participants in Cohort 2 had SRI on HD and mild-to-moderate COVID-19 disease with confirmed SARS-CoV-2 infection and initial onset of signs/symptoms attributable to COVID-19 within 5 days prior to the day of treatment assignment. All eligible participants were assigned to receive a single dose of PF-07321332 (nirmatrelvir)/ritonavir 300 mg/100 mg orally on Day 1 followed by PF-07321332 (nirmatrelvir)/ritonavir 150 mg/100 mg QD from Day 2 to Day 5.
Period: Overall Study
Arm/Group | Cohort 1 (No HD) | Cohort 2 (Intermittent HD)
Started | 3 | 12
Completed | 3 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline population was the safety analysis set (SAS) which was all participants enrolled and took at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (No HD) | Cohort 2 (Intermittent HD) | Total
Number analyzed (Participants) | 3 | 12 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (29.10) | 52.8 (13.24) | 54.7 (16.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 8
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 1 | 8 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 3 | 8 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious AEs (SAEs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was defined as any untoward medical occurrence that, at any dose, meets one or more of the following criteria: 1. results in death. 2. is life-threatening. 3. Requires inpatient hospitalization or prolongation of existing hospitalization. 4. Results in persistent or significant disability/incapacity. 5. Is a congenital anomaly/birth defect. 6. Is a suspected transmission via a Pfizer product of an infectious agent, pathogenic or nonpathogenic. 7. other important medical events. Any events occurring following start of treatment were considered treatment emergent.
Time Frame: From start of treatment on Day 1 to Day 34
Population: The analysis population was the SAS which was all participants assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (No HD) | Cohort 2 (Intermittent HD)
Number analyzed (Participants) | 3 | 12
Participants
  Participants with treatment emergent AEs | 1 | 2
  Participants with treatment emergent SAEs | 0 | 1

2. Primary Outcome: Number of Participants With Permanent Discontinuation From Study or Study Intervention Due to Adverse Events and Serious Adverse Events
Description: as for outcome 1
Time Frame: From start of treatment on Day 1 to Day 34
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (No HD) | Cohort 2 (Intermittent HD)
Number analyzed (Participants) | 3 | 12
Participants
  Permanent Discontinuation From Study | 0 | 0
  Permanent Discontinuation From Study Intervention | 0 | 1

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of PF-07321332 (Nirmatrelvir)
Description: Nirmatrelvir plasma concentration data were analyzed using nonlinear mixed effects models. Time frame was: For Cohort 1: Day 1 (anytime between 1-3 hours post-dose), Day 2 (anytime between 4-8 hours post-dose), Day 3 (anytime between 9-15 hours post-dose), Day 4 (pre-dose, anytime between 1-4 hours post-dose), Day 5 (pre-dose, anytime between 0.5-6 hours post-dose, anytime between 9-15 hours post-dose). For Cohort 2: Day 1 (anytime between 1-3 hours post-dose), Day 3 (pre-HD), Day 4 (pre-HD, pre-dose, anytime between 0.5-3 hours post-dose, anytime between 4-8 hours post-dose, anytime between 9-15 hours post-dose).
Time Frame: Treatment Day 1 to Day 5, see description for details
Population: All participants assigned to study intervention and treated who had at least 1 PK parameter measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1 (No HD) | Cohort 2 (Intermittent HD)
Number analyzed (Participants) | 2 | 12
nanogram per milliliter (ng/mL) | NA (NA) — There were only 2 participants with evaluable data. Per the Sponsor's clinical pharmacology rule book, only minimum and maximum values were presented for a parameter with less than 3 evaluable measurements. The minimum value was 3040 ng/mL and the maximum value was 5600 ng/mL. | 3280 (48)

4. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Nirmatrelvir
Description: Vz/F was estimated at steady state.
Time Frame: Treatment Day 1 to Day 5
Population: All participants assigned to study intervention and treated who had at least 1 PK parameter measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Cohort 1 (No HD) | Cohort 2 (Intermittent HD)
Number analyzed (Participants) | 2 | 12
Liter (L) | NA (NA) — There were only 2 participants with evaluable data. Per the Sponsor's clinical pharmacology rule book, only minimum and maximum values were presented for a parameter with less than 3 evaluable measurements. The minimum value was 79.2 L and the maximum value was 73.3 L. | 99.8 (49)

5. Primary Outcome: Area Under the Curve Over a Dosing Interval (AUC0-tau) of Nirmatrelvir
Description: AUC0-tau was measured at 24 hours post-dose.
Time Frame: 24 Hours after each dose on Treatment Day 1 to Day 5
Population: All participants assigned to investigational product and treated who had at least 1 PK parameter measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Cohort 1 (No HD) | Cohort 2 (Intermittent HD)
Number analyzed (Participants) | 2 | 12
nanogram*hour per milliliter (ng*hr/mL) | NA (NA) — There were only 2 participants with evaluable data. Per the Sponsor's clinical pharmacology rule book, only minimum and maximum values were presented for a parameter with less than 3 evaluable measurements. The minimum value was 69800 ng*hr/mL and the maximum value was 131000 ng*hr/mL. | 65740 (59)

6. Primary Outcome: Terminal Half-Life (T1/2) of Nirmatrelvir
Description: T1/2 was observed directly from data.
Time Frame: Treatment Day 1 to Day 5
Population: All participants assigned to study intervention and treated who had at least 1 of PK parameter measured.
Measure: Mean (Standard Deviation); unit: Hour (hr)
Arm/Group | Cohort 1 (No HD) | Cohort 2 (Intermittent HD)
Number analyzed (Participants) | 2 | 12
Hour (hr) | NA (NA) — There were only 2 participants with evaluable data. Per the Sponsor's clinical pharmacology rule book, only minimum and maximum values were presented for a parameter with less than 3 evaluable measurements. The minimum value was 45.7 hr and the maximum value was 102 hr. | 78.93 (49.761)

7. Primary Outcome: Trough Concentration (Ctrough) of Nirmatrelvir
Description: Ctrough was measured at 24 hours post-dose (pre the next dose). It was analyzed using nonlinear mixed effect models.
Time Frame: 24 Hours after each dose on Treatment Day 1 to Day 5
Population: All participants assigned to study intervention and treated who had at least 1 PK parameter measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 (No HD) | Cohort 2 (Intermittent HD)
Number analyzed (Participants) | 2 | 12
ng/mL | NA (NA) — There were only 2 participants with evaluable data. Per the Sponsor's clinical pharmacology rule book, only minimum and maximum values were presented for a parameter with less than 3 evaluable measurements. The minimum value was 2720 ng/mL and the maximum value was 5490 ng/mL. | 2188 (81)

8. Secondary Outcome: Hemodialysis Clearance (CLd) of Nirmatrelvir
Description: CLd of nirmatrelvir was calculated for Cohort 2 using non-compartmental analysis of arterial and venous port plasma concentration-time data. Only participants in Cohort 2 were on hemodialysis.
Time Frame: Pre-dose, 0.5, 1, 2, 3 and 4 hours post-dose on Day 3 and Day 4
Population: All participants assigned to study intervention and treated who had at least 1 of the PK parameters of interest measured. Here, overall number of participants analyzed signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per minute (mL/min)
Arm/Group | Cohort 2 (Intermittent HD)
Number analyzed (Participants) | 11
milliliter per minute (mL/min) | 30.53 (35)

9. Secondary Outcome: Fraction of Drug Removed During Dialysis (Fd) of Nirmatrelvir
Description: Fd of nirmatrelvir was calculated for Cohort 2 using non-compartmental analysis of arterial and venous port plasma concentration-time data. Only participants in Cohort 2 were on hemodialysis.
Time Frame: Pre-dose, 0.5, 1, 2, 3 and 4 hours post-dose on Day 3 and Day 4
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of drug removed
Arm/Group | Cohort 2 (Intermittent HD)
Number analyzed (Participants) | 11
Percentage of drug removed | 6.937 (138)

ADVERSE EVENTS:
Time Frame: From start of treatment on Day 1 to Day 34
Arm/Group | Cohort 1 (No HD) | Cohort 2 (Intermittent HD)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/12
Other Adverse Events (participants affected / at risk) | 1/3 | 2/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (No HD) (N=3) | Cohort 2 (Intermittent HD) (N=12)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Hypertensive nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (No HD) (N=3) | Cohort 2 (Intermittent HD) (N=12)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Brain natriuretic peptide increased (Investigations) | 0 | 1
Headache (Nervous system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclosure previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT05487040/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT05487040/SAP_001.pdf